CLINICAL TRIAL: NCT03452683
Title: The Use of a Symptom and Weight e-Diary Among Patients With Heart Failure
Brief Title: e-Diary in Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Competing trials
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Linda Park, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: e-Diary in Heart Failure
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants randomized to the Usual Care arm will receive educational handouts.
- Movn Mobile App (Experimental): Participants randomized to the Movn Mobile App arm will have the Movn app downloaded to their cell phone. Participants will enter in their weight and symptoms into the app every day.
  Interventions: Behavioral: Movn Mobile App

INTERVENTIONS:
Behavioral: Movn Mobile App — Movn is a mobile application that is downloaded to a cell phone where participants can enter their weight and symptoms every day.
  Arms: Movn Mobile App

SUMMARY:
The purpose of this study is to determine the efficacy and feasibility of using a smartphone application to monitor symptoms and weight in patients with advanced heart failure.

DETAILED DESCRIPTION:
Attention to symptoms of heart failure and weight gain are central tenets in heart failure patient education and self-care. A key self-care skill for heart failure patients is the early detection of subtle changes in symptoms. Daily diary use can be one method for patients to acknowledge and attend to their symptoms. This study is examining if the use of a diary in the form of an app on a mobile phone will improve patient outcomes. Participants will be randomized to one of two groups-- usual care or the Movn mobile application. Participants randomized to the mobile app will be asked to record their weight and any symptoms every day over the course of two months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* History of symptomatic heart failure (Class III or IV)
* Owns a smartphone or tablet compatible with the Movn mobile application

Exclusion Criteria:

* Cognitive impairment
* Lack of English proficiency/literacy
* Clinically unstable (decompensated heart failure NYHA class 3-4; unstable arrhythmias, aortic stenosis, thrombophlebitis, dissecting aneurysm, or symptomatic anemia; active infection; uncontrolled blood pressure: resting diastolic higher than 100 mmHg, systolic greater than 180 mmHg; unstable angina, 2nd or 3rd degree heart block; or uncontrolled high grade exercise-induced ventricular ectopy or hemodynamically unstable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Health Care Utilization | Health Care Utilization will be measured at two timepoints-- baseline and month 3.
  Health Care Utilization will be measured by a questionnaire that asks about number of office visits, emergency room visits, and hospitalization in the last 60 days.

SECONDARY OUTCOMES:
Quality of Life | Quality of life will be measured at two timepoints-- baseline and month 3.
  Quality of life will be measured by the 20-item Short Form Survey (SF-20). Scores range from 0 to 100 with high values indicating higher functioning.
Depression | Depression will be measured at baseline and month 3.
  Depression will be measured by the Patient Health Questionnaire (PHQ-9). Scores can range from 5 to greater than 20 with 5 indicating minimal symptoms and 20 indicating severe major depression.
Satisfaction with the app | Satisfaction with the app will be measured at month 3.
  Participation satisfaction with the mobile app will be assessed through individual interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- John Muir Medical Center, Concord, California, United States

IPD SHARING:
Plan to Share IPD: Undecided